CLINICAL TRIAL: NCT05577598
Title: Glucose Consumption During Deep Brain Stimulation With Functional [18F]FDG-Brain-PET in Obsessive-Compulsive Disorder
Acronym: OCDBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christoph Kraus, Ap. Prof. PD, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: V4 03062020
Record Dates: First submitted 2022-09-25; First posted 2022-10-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Obsessive-Compulsive Disorder; Psychiatric Disorder
Keywords: FDG-PET; Deep Brain Stimulation; Brain Glucose Consumption
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Mental Disorders

STUDY DESIGN:
Intervention Model Description: After 8 weeks of open label DBS optimization and treatment, randomization to 12 weeks active or 12 weeks sham DBS treatment followed by a crossover switch at study week 24 to the opposing condition.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Subjects in this arm will receive active stimulation. (Active Comparator): The Medtronic DBS system will be implanted in subjects in both study arms. Stimulation will vary depending on the study arm assignment. All subjects will receive therapeutic settings at the end of the blinded period.
  Interventions: Device: Implantation of a DBS therapy system
- Subjects in this arm will receive sham stimulation with DBS being turned off. (Sham Comparator): The Medtronic DBS system will be implanted in subjects in both study arms. Stimulation will vary depending on the study arm assignment. All subjects will receive therapeutic settings at the end of the blinded period.
  Interventions: Device: Implantation of a DBS therapy system

INTERVENTIONS:
Device: Implantation of a DBS therapy system — The system is called "Reclaim DBS Therapy for OCD" und is marketed by Medtronic (Minneapolis, Minnesota). It has a HDE status by the FDA. The system consists of two quadripolar electrodes (Medtronic Reclaim DBS) as well as a generator (Medtronic Activa PC), which will be implanted into a subcutaneous pocket below the clavicula.

SUMMARY:
The purpose of this randomized, sham-controlled study is to evaluate the effectiveness of DBS therapy in individuals suffering from severe OCD and to investigate DBS treatment with functional [18F]FDG-Brain-PET.

DETAILED DESCRIPTION:
The overall planned study duration per subject is 36 weeks, whereby inclusion is timepoint zero and implantation of DBS will be conducted during the first four study weeks. Patients will then undergo an 8-week open-label active DBS treatment phase followed by a 12-week double blind active or sham treatment and finally a 12-week crossover period with the inverse (active/sham) treatment with at least biweekly study visits. Patients as well as patient handling study psychiatrists will be blinded to active/sham. In case of unbearable aggravation of the symptoms during sham, the sham-period will be shortened to a tolerable length. After maximal 38 weeks all study procedures will be completed, and active DBS treatment will be maintained as long as clinically necessary.

ELIGIBILITY:
Inclusion Criteria:

* a score of 25 or higher on the Yale-Brown Obsessive Compulsive Scale
* previous failure to respond to at least two medication trials with serotonin reuptake inhibitors at or, if tolerated, beyond the FDA maximum recommended dose for a minimum duration over at least ten weeks each.
* at least one trial with tricyclic medication at or, if tolerated, beyond the FDA maximum recommended dose for a minimum duration over at least ten weeks each.
* at least one trial of augmentation with antipsychotic medication, lithium, a benzodiazepine or buspirone
* at least on trial of psychotherapy (cognitive behavioral therapy or comparable techniques) for at least 20 sessions
* ability to provide written informed consent

Exclusion Criteria:

* any history of current or past psychotic disorder
* a manic episode within the preceding three years
* any current clinically significant medical or neurological disorder, that is a contraindication against DBS
* any disease that could lead to an altered glucose reactivity (e.g. diabetes)
* any clinically significant preoperative MRI abnormality or inability to undergo presurgical MRI
* current or unstable remitted substance abuse or dependence except nicotine
* pregnancy or high risk of becoming pregnant during study duration (desire to have children) and refusal to utilize a proper method of contraception
* Any current severe personality disorder except comorbid anankastic personality disorder
* Inability to follow the study protocol or adhere to operational requirements
* Current and unstable suicidality

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of metabolic rates of glucose response pattern | fPET measurements will take place in Week 4 and Week 5 of the trial.
  Change of metabolic rates of glucose response pattern

SECONDARY OUTCOMES:
Determination of association between metabolic (change in glucose consumption - PET), structural (white matter pathways - DTI) and functional connectivity (resting state fMRI - functional connectivity patterns) | Data acquisition will take place during screening and in the first 5 weeks of the study.
  Combination of [18F]FDG-PET data with DTI and resting state fMRI data
Change in YBOCS scores by active DBS treatment and sham treatment | Week 1 to 38
  Comparison of YBOCS scores during active and sham treatment
Correlation of metabolic (change in glucose consumption) and connectivity measures (white matter pathways) with clinical outcomes (YBOCS) and neuropsychological tests (SSRT, n-back, WCST) | Data acquisition will take place during screening and in Week 1 to Week 38 of the study.
  YBOCS will serve as a marker for clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kraus, MD PhD, Principal Investigator — Medical University of Vienna, Department of Psychiatry and Psychotherapy
Locations (1):
- Medical University of Vienna, Department of Psychiatry and Psychotherapy, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No